CLINICAL TRIAL: NCT05636969
Title: Effects of Multimodal Prehabilitation on Cardiorespiratory Fitness and Pulmonary Function During Neoadjuvant Therapy in Patients with Locally Advanced Lung Cancer
Brief Title: Multimodal Prehabilitation in Patients with Lung Cancer Undergoing Neoadjuvant Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundació Sanitaria de Mollet (Unknown); Hospital General de Granollers (Unknown); Consorci Hospitalari de Vic (Other); CHU de Rouen - Accueil (Other)
Responsible Party: Principal Investigator, Graciela Martinez-Palli, Senior Consultant, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCB-TNA-2022
Record Dates: First submitted 2022-11-20; First posted 2022-12-05 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to whether patients receiving prehabilitation or not for some outcome measures (complications, neoadjuvant-related outcomes). Researchers conducting analyses will be blinded to patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prehabilitation (Experimental): Patients in this group will attend a supervised multimodal prehabilitation programme
  Interventions: Behavioral: Multimodal prehabilitation
- Control (No Intervention): Patients declining participation in the prehabilitation program will serve as controls and will receive standard recommendations to increase or maintain their physical activity levels and fitness during the neoadjuvant therapy

INTERVENTIONS:
Behavioral: Multimodal prehabilitation — The multimodal prehabilitation programme will consist of 1) twice weekly, supervised exercise training at the hospital gym for approximately 12-16 weeks; 2) nutritional consultation and diet optimization and supplementation if needed; 3) individual or group-based psychological support.
  Arms: Prehabilitation

SUMMARY:
Neoadjuvant therapy (NAT) with chemoimmunotherapy is currently indicated for patients with locoregional advanced non-small cell lung cancer (NSCLC) prior to resection surgery, but literature has suggested that this is associated with decreased pulmonary function and potentially cardiorespiratory fitness, leading to increased risk of postoperative complications. In this study, we aimed to: 1) compare the effects of NAT on cardiorespiratory fitness (VO2peak) and lung function (DLCO, FEV1 and FVC) in patients with locoregional lung cancer undergoing prehabilitation before lung resection surgery.

Secondary objectives included:

1. To determine feasibility of the intervention (recruitment rate, competition rate and adherence) as well as safety (incidence of adverse events), particularly regarding the exercise component;
2. To quantify the effects of the intervention in terms of functional capacity (1min Sit-to-Stand Test), mood (Hospital Anxiety and Depression Scale) and self-reported physical activity (Yale Physical Activity Survey).
3. To assess the effects of multimodal prehabilitation on treatment completion (dose reductions/delays in planning/treatment withdrawal) as well as tolerability/toxicity (Coming Terminology Criteria for Adverse Events version 4.03) to chemo/immunotherapy
4. To assess the effects of multimodal prehabilitation on surgical outcomes (postoperative complications based on the Comprehensive Complication Index (CCI) of the Clavien-Dindo Classification System and length of hospital stay).
5. To determine the effect of the intervention on post-operative functional recovery by means of the 1-min Sit-To-Stand test conducted at hospital discharge.

In order to achieve this, we will conduct a prospective study including all patients with NSCLC scheduled for NAT (chemoimmunotherapy or chemotherapy alone) across four different hospitals in Spain and France. Patients will be identified from the multidisciplinary tumour board and will be subsequently referred to the oncologist consultation. After this, one of the members of the researchers will contact the patient and explain the purpose of the study. Those who are willing to participate, will be scheduled to undergo a CardioPulmonary Exercise Test (CPET) in addition to standard lung function tests (spirometry, diffusion capacity of carbon monoxide). After that, patients will be invited to participate in a multimodal prehabilitation program including supervised exercise training, home-based inspiratory muscle training, nutritional optimization and psychological support. Patients who refuse participation in the program due to logistic reasons, will be asked to serve as controls. In addition, we will also use data from a historical cohort including patients treated with chemoimmunotherapy prior to the implementation of the study as controls.

Patients will be assessed at baseline, after NAT and post-surgery (at hospital discharge).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with diagnosed non-small celll lung cancer (NSCLC) undergoing neoadjuvant therapy before lung resection surgery

Exclusion Criteria:

* Physical impairments that prevent patients to perform a CardioPulmonary Exercise Test
* Non-resectable tumours
* Patients who refuse either surgical resection or neoadjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in cardiorespiratory fitness assessed with a cardiopulmonary exercise test | 2 weeks post-neoadjuvant therapy
  Differences in maximum oxygen consumption (VO2pic) pre to post neoadjvuant therapy during an incremental, symptom-limited test

SECONDARY OUTCOMES:
Changes in diffusion capacity of carbon monoxide (DLCO) | 2 weeks post-neoadjuvant therapy
  Differences in diffusion capacity of carbon monoxide pre to post-neoadjuvant therapy
Changes in submaximal cardiorespiratory fitness assessed with a cardiopulmonary exercise test | 2 weeks post-neoadjuvant therapy
  Differences in oxygen consumption at the anaerobic threshold (VO2AT) pre to post-neoadjuvant therapy during an incremental, symptom-limited test
Changes in ventilatory efficiency (VE/VCO2 slope) assessed during a cardiopulmonary exercise test | 2 weeks post-neoadjuvant therapy
  Changes in ventilatory efficiency (VE/VCO2 slope) pre to post-neoadjuvant therapy
Changes in pulmonary function (FEV1) | 2 weeks post-neoadjuvant therapy
  Differences observed in the maximum volume achieved during the first second (FEV1) of a forced spirometry test, pre to post-neoadjuvant therapy
Changes in pulmonary function (FVC) | 2 weeks post-neoadjuvant therapy
  Differences observed in the forced ventilatory capacity (FVC) of a forced spirometry test, pre to post-neoadjuvant therapy
Feasibility (recruitment rate ) of multimodal prehabilitation | 1 week before surgery
  Feasibility of the multimodal prehabilitation programme assessed by the recruitment rate (number of patients attending prehabilitation versus number of eligible patients)
Feasibility (completion rate) of multimodal prehabilitation | 1 week before surgery
  Feasibility of the multimodal prehabilitation programme assessed by the completion rate (number of completers among those who accepted to participate in the programme)
Adherence | 1 week before surgery
  Number of completed exercise sessions in the prehabilitation cohort versus number of scheduled sessions
Adverse events | 1 week before surgery
  Number of adverse events registered during the exercise training sessions
Postoperative Complications | within 30 days of hospital discharge
  Number and severity of postoperative complications will be assessed by reviewing medical records and calculating the Comprehensive Complication Index (CCI) according to the Clavien-Dindo Classification.
30-Day readmissions, re-interventions and emergency room visits | 30 days after surgery
  Readmissions, surgical re-interventions and emergency room visits post-discharge and during the first 30 days will be recorded by reviewing medical records
Chemoimmunotherapy completion rates | 1 week post-neoadjuvant therapy
  Chemoimmunotherapy complete dosage, treatment delays and treatment withdrawal rates will be calculated and compared in both groups
Post-surgery functional capacity | Same day as dicharge from hospital
  Functional capacity assessed with the 1 min Sit-to-Stand Test which consist of counting the number of times the patient can stand up and sit back onto a chair without arm support during one minute.
Post-NAT functional capacity | 2 weeks post-neoadjuvant therapy
  Functional capacity assessed with the 1 min Sit-to-Stand Test which consist of counting the number of times the patient can stand up and sit back onto a chair without arm support during one minute.
Post-NAT mood | 2 weeks post-neoadjuvant therapy
  Anxiety and depression symptoms will be assessed with a self-administer questionnaire, the Hospital Anxiety and Depression Scale
Post-NAT self-reported physical activity | 2 weeks post-neoadjuvant therapy
  Self-reported physical activity levels will be measured using a validated questionnaire, the Yale Physical Activity Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunelli A, Rocco G, Szanto Z, Thomas P, Falcoz PE. Morbidity and mortality of lobectomy or pneumonectomy after neoadjuvant treatment: an analysis from the ESTS database. Eur J Cardiothorac Surg. 2020 Apr 1;57(4):740-746. doi: 10.1093/ejcts/ezz287. PMID 31638692
- [Background] Cabanero Sanchez A, Munoz Molina GM, Fra Fernandez S, Muriel Garcia A, Cilleruelo Ramos A, Martinez Hernandez N, Hernando Trancho F, Moreno Mata N; GE-VATS. Impact of neoadjuvant therapy on postoperative complications in non-small-cell lung cancer patients subjected to anatomic lung resection. Eur J Surg Oncol. 2022 Sep;48(9):1947-1953. doi: 10.1016/j.ejso.2022.03.008. Epub 2022 Mar 29. PMID 35379545
- [Background] Connolly JG, Fiasconaro M, Tan KS, Cirelli MA Jr, Jones GD, Caso R, Mansour DE, Dycoco J, No JS, Molena D, Isbell JM, Park BJ, Bott MJ, Jones DR, Rocco G. Postinduction therapy pulmonary function retesting is necessary before surgical resection for non-small cell lung cancer. J Thorac Cardiovasc Surg. 2022 Aug;164(2):389-397.e7. doi: 10.1016/j.jtcvs.2021.12.030. Epub 2021 Dec 23. PMID 35086669
- [Background] Jack S, West MA, Raw D, Marwood S, Ambler G, Cope TM, Shrotri M, Sturgess RP, Calverley PM, Ottensmeier CH, Grocott MP. The effect of neoadjuvant chemotherapy on physical fitness and survival in patients undergoing oesophagogastric cancer surgery. Eur J Surg Oncol. 2014 Oct;40(10):1313-20. doi: 10.1016/j.ejso.2014.03.010. Epub 2014 Mar 27. PMID 24731268
- [Background] Sinclair R, Navidi M, Griffin SM, Sumpter K. The impact of neoadjuvant chemotherapy on cardiopulmonary physical fitness in gastro-oesophageal adenocarcinoma. Ann R Coll Surg Engl. 2016 Jul;98(6):396-400. doi: 10.1308/rcsann.2016.0135. Epub 2016 May 3. PMID 27138851
- [Background] Silver JK, Baima J. Cancer prehabilitation: an opportunity to decrease treatment-related morbidity, increase cancer treatment options, and improve physical and psychological health outcomes. Am J Phys Med Rehabil. 2013 Aug;92(8):715-27. doi: 10.1097/PHM.0b013e31829b4afe. PMID 23756434
- [Background] Granger C, Cavalheri V. Preoperative exercise training for people with non-small cell lung cancer. Cochrane Database Syst Rev. 2022 Sep 28;9(9):CD012020. doi: 10.1002/14651858.CD012020.pub3. PMID 36170564
- [Background] Allen SK, Brown V, White D, King D, Hunt J, Wainwright J, Emery A, Hodge E, Kehinde A, Prabhu P, Rockall TA, Preston SR, Sultan J. Multimodal Prehabilitation During Neoadjuvant Therapy Prior to Esophagogastric Cancer Resection: Effect on Cardiopulmonary Exercise Test Performance, Muscle Mass and Quality of Life-A Pilot Randomized Clinical Trial. Ann Surg Oncol. 2022 Mar;29(3):1839-1850. doi: 10.1245/s10434-021-11002-0. Epub 2021 Nov 1. PMID 34725764
- [Derived] Chen YX, Sebio-Garcia R, Arguis MJ, Reguart N, Arcocha A, Navarro A, Navarro-Ripoll R, Boujibar F, Munoz-Borrajo S, Boada M, Urena A, Guirao A, Siso M, Cardena-Gutierrez A, Perez-Garcia R, Bello I, Martinez-Palli G. Multimodal prehabilitation to prevent loss of cardiorespiratory fitness in patients with locally advanced lung cancer undergoing chemoimmunotherapy: protocol for a non-randomized multicentre study. Transl Lung Cancer Res. 2025 Sep 30;14(9):4057-4067. doi: 10.21037/tlcr-2025-311. Epub 2025 Sep 28. PMID 41133003